CLINICAL TRIAL: NCT00779363
Title: A Prospective Clinical Trial of the TANTALUS System In Treatment of Obese to Morbidly Obese Patients
Brief Title: A Prospective, Clinical Trial of the TANTALUS® System in Treatment of Obese to Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaCure (USA), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC CR TAN2007-012
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: obese,; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implanted Device (Experimental)
  Interventions: Device: rechargeable TANTALUS II

INTERVENTIONS:
Device: rechargeable TANTALUS II — Subjects will undergo an approximately two week baseline screening process. Eligible subjects will undergo device implantation. This will be followed by therapy initiation approximately one week after implantation. The device will then be activated to automatically deliver gastric contractility modulating (GCM) for 12 weeks of therapy. Stimulation will continue in for a safety monitoring period of 18 months following the therapy period.

SUMMARY:
The objectives of this feasibility study are to evaluate the safety and functionality of the TANTALUS System with TANTALUS II IPG, to assess the effect of GCM signal application on trends of HbA1c, blood glucose and body weight changes.

DETAILED DESCRIPTION:
This is a prospective multi center, non-randomized, treatment only clinical trial with up to thirty (30) obese with type 2 diabetes subjects. The study is designed to demonstrate that use of the rechargeable TANTALUS II IPG is safe and that it functions as designed.

Subjects will undergo an approximately two week baseline screening process. Eligible subjects will undergo device implantation. This will be followed by therapy initiation approximately one week after implantation. The device will then be activated to automatically deliver gastric contractility modulating (GCM) for 12 weeks of therapy. Stimulation will continue in for a safety monitoring period of 18 months following the therapy period.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70 years
* Diabetic subjects having HbA1c greater than or equal to 7.5% and less than or equal to 9.5 % at Visit 1
* Sex: male or female. Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.
* Type 2 diabetes duration less than 10 years but at least 6 months
* Type 2 diabetic Subjects taking no more than two (2) oral anti-diabetic agents [Sulfonylurea, Metformin or thiazolinedione (TZD)].
* Stable anti-diabetic drugs for at least three (3) months prior to enrollment and six (6) months for thiazolinedione (TZD).
* Fasting blood glucose values > 120 and < 240 mg/dl at baseline
* Stable HbA1c, described as no significant change (≤ 0.5% variation) between a historical value in the subjects' medical record within 3 months prior to enrollment and the A1c value gathered at baseline.
* If subject is under anti-depressant medication, the treatment needs to be stable for at least six (6) months prior to enrollment.
* BMI between 28 and 45 (kg/m2)
* Stable weight, defined as no significant weight change over the three months prior to enrollment as reported by the subject (±5 kg).
* Stable medications (including anti-hypertensive and lipid-lowering) for at least one month prior to enrollment.
* Compliant, willing and able to participate in the follow-up visits for the study duration.
* Alert, mentally competent, and able to understand and comply with the requirements of the clinical trial, and personally motivated to abide by the requirements and restrictions of the clinical trial.
* Able to provide voluntary informed consent.

Exclusion Criteria:

* Gastroparesis or intestinal pseudo-obstruction.
* Receiving medications known to affect gastric motility.
* Taking appetite suppressant or weight loss medications within 1 month of enrollment.
* Diabetic subjects on insulin.
* Past or current psychiatric condition that may impair his or her ability to comply with the study procedures.
* Severe eating disorders such as bulimia or binge eating.
* Obese due to a clinically diagnosed endocrine problem.
* Pregnant (proven by positive βhCG), or lactating.
* History of anemia (<10 g/dl) over past 3-months.
* Prior bariatric surgery.
* History of peptic ulcer disease.
* Use of another investigational device or agent in the 30 days prior to enrollment.
* Participation in another clinical study.
* Life threatening co-morbidity or life expectancy of less than one year.
* Myocardial Infarction or one or more episodes of unstable angina within six months prior to enrollment.
* Implanted with a permanent pacemaker, an automatic implantable defibrillator, or other electro-stimulation device.
* History of life threatening disease within 5 years of enrollment.
* Use of routine ulcerogenic drugs.
* Use of prescription, over the counter or herbal weight loss products.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation | June 2004-September2009
Device Functionality Evaluation | June 2004-September2009

SECONDARY OUTCOMES:
Change in HbA1c | June 2004-September2009
Percentage of body weight loss | June 2004-September2009

CONTACTS AND LOCATIONS:
Overall Officials: Harold Lebowitz, MD, Study Chair — Proffesor of Medicine, Endocrinology and Metabolism/Diabetes, State University on NY Health Science
Locations (2):
- United States (2):
  - Cedars Sinai, Los Angeles, California
  - Diabetes and Glandular Disease Clinic (DGD), San Antonio, Texas